CLINICAL TRIAL: NCT00626925
Title: Topiramate Treatment of Problem Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Henry Kranzler, Professor of Psychiatry, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-052-2; P60AA003510 (NIH); M01RR006192 (NIH)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Alcohol Drinking
Keywords: Randomized Trial; Medication for Heavy Drinking; Topiramate Treatment
MeSH Terms: conditions — Alcohol Drinking | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Topiramate Group (Active Comparator): topiramate capsules beginning at 25 mg/day with gradual increase to a maximum of 200 mg orally)
  Interventions: Drug: topiramate
- Total Placebo Group (Placebo Comparator): inactive placebo matched in appearance with topiramate capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: topiramate — up to 200mg/day orally (over 12 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
  Other Names: Topamax
  Arms: Total Topiramate Group
Drug: placebo — placebo (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
  Arms: Total Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of topiramate in reducing drinking and heavy drinking frequency in problem drinkers. We hypothesize that at a dosage of up to 200mg/day, topiramate will be well tolerated in this patient population and that, compared to placebo treatment, topiramate will result in a greater reduction in the frequency of both drinking days and heavy drinking days.

DETAILED DESCRIPTION:
It is estimated that 30% of the general population are problem drinkers (NIAAA 2007). Despite its high prevalence, problem drinkers are understudied, particularly with respect to medications that may help them to reduce their drinking to safe levels. The study will extend to this patient population findings from a trial of topiramate, which showed the drug to be well tolerated and efficacious in moderately-severe alcohol-dependent patients (Johnson et al. 2003).

This is a 13-week, double-blind, placebo-controlled study of topiramate (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper) and medical management counseling to reduce drinking among problem drinkers (i.e., heavy drinkers without evidence of physical dependence on alcohol) who want to reduce their drinking.

Participants attend weekly study visits for the first 5 weeks and then bi-weekly visits for the last 8 weeks of the study, and are randomly assigned to receive topiramate or placebo on a daily basis. In addition to study visits, participants report daily moods, drinking, and medication usage through an Interactive Voice Response (IVR) system they call each night. In-person follow-up evaluations are conducted at 3 and 6 months post-treatment to provide a measure of the durability of treatment effects. This study also aims to examine the relation between genotype and the response to topiramate treatment.

An additional aim is to conduct a substudy to examine neural cells generated from skin fibroblast cells obtained from study participants via a skin biopsy (participation in the substudy is completely optional). Initially, we will examine variables key to reliably generating neurons from the cells and characterize these neurons using a variety of laboratory measures. A longer term goal is to compare gene expression in individuals who show a robust reduction in drinking following treatment with topiramate with those who show no beneficial treatment effects.

A second additional aim is to explore whether the therapeutic and adverse effects of topiramate are similar in patients on a stable regimen of an antidepressant to those not receiving such therapy. Although exploratory, given the absence of data that directly address this issue, we will stratify subjects by the presence or absence of current antidepressant therapy.

Careful evaluation of the study's hypotheses will provide important information on the efficacy and mechanism of effects of topiramate as a treatment for problem drinkers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years, inclusive;
* have an average weekly ethanol consumption of >=24 standard drinks for men, or >=18 standard drinks for women;
* be able to read English at the 8th grade or higher level and show no evidence of significant cognitive impairment;
* be willing to nominate an individual who will know the patient's whereabouts in order to facilitate follow up during the study;
* if a woman of child-bearing potential (i.e., who has not had a hysterectomy, bilateral oophorectomy, tubal ligation or who are less than two years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment;
* if applicable, individuals being treated with a single antidepressant that has been stable in dosage for a minimum of four weeks; and
* be willing to provide signed, informed consent to participate in the study (including a willingness to reduce drinking to non-hazardous levels).

Exclusion Criteria:

* a current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including direct bilirubin elevations of >110% or transaminase elevations >300% normal (We will not exclude patients with hypertension, diabetes mellitus, asthma or other common medical conditions, as long as these are adequately controlled and the patient has an ongoing relationship with a primary-care practitioner);
* a history of nephrolithiasis;
* a history of glaucoma;
* a serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, panic disorder, borderline or antisocial personality disorder, organic mood or mental disorders, eating disorder, or substantial suicide or violence risk) on the basis of history or psychiatric examination;
* a current Diagnostic & Statistical Manual of Mental Disorders 4th ed (DSM-IV) diagnosis of drug dependence (other than nicotine dependence);
* a current Diagnostic and Statistical Manual of Mental Disorders 4th ed (DSM-IV) diagnosis of alcohol dependence that is clinically moderate or severe;
* a history of hypersensitivity to topiramate;
* currently taking any tricyclic antidepressant (e.g., Adapin (doxepin), Anafranil (clomipramine), Elavil (amitryptyline), Pamelor (nortryptyline), Tofranil (imipramine), Sinequan (doxepin); or
* are considered by the investigators to be an unsuitable candidate for receipt of an investigational drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Kranzler, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kranzler HR, Feinn R, Pond T, Hartwell E, Gelernter J, Crist RC, Witkiewitz K. Post-treatment effects of topiramate on alcohol-related outcomes: A combined analysis of two placebo-controlled trials. Addict Biol. 2022 Mar;27(2):e13130. doi: 10.1111/adb.13130. PMID 35229945
- [Derived] Kranzler HR, Hartwell EE, Feinn R, Pond T, Witkiewitz K, Gelernter J, Crist RC. Combined analysis of the moderating effect of a GRIK1 polymorphism on the effects of topiramate for treating alcohol use disorder. Drug Alcohol Depend. 2021 Aug 1;225:108762. doi: 10.1016/j.drugalcdep.2021.108762. Epub 2021 May 21. PMID 34049101
- [Derived] Feinn R, Curtis B, Kranzler HR. Balancing risk and benefit in heavy drinkers treated with topiramate: implications for personalized care. J Clin Psychiatry. 2016 Mar;77(3):e278-82. doi: 10.4088/JCP.15m10053. PMID 26891181
- [Derived] Kranzler HR, Armeli S, Feinn R, Tennen H, Gelernter J, Covault J. GRIK1 genotype moderates topiramate's effects on daily drinking level, expectations of alcohol's positive effects and desire to drink. Int J Neuropsychopharmacol. 2014 Oct;17(10):1549-56. doi: 10.1017/S1461145714000510. Epub 2014 Apr 30. PMID 24786948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated at the University of Connecticut Health Center in March 2008 and was transferred to the University of Pennsylvania in December 2010. The last study visit was completed on 11/20/2013. We enrolled a total of 200 subjects, randomizing 138 to study medication. We recruited participants using flyers, newspaper and radio ads.
Groups:
- Active Med: topiramate (up to 200 mg orally)
  topiramate: up to 200mg/day orally (over 12 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
- Placebo: placebo
  placebo: placebo (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
Period: Overall Study
Arm/Group | Active Med | Placebo
Started | 67 | 71
Completed | 55 | 62
Not Completed | 12 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — relapse | 1 | 0
Not completed — Adverse effect | 6 | 2
Not completed — Lack of Efficacy | 1 | 4
Not completed — Time constraints | 3 | 1

BASELINE CHARACTERISTICS:
Population: In the Total topiramate and Placebo group e included all subjects enrolled who were randomized into the study based.
Groups:
- Total Topiramate Group: topiramate (up to 200 mg orally)
  topiramate: up to 200mg/day orally (over 12 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
- Total Placebo Group: placebo
  placebo: placebo (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
- Total: Total of all reporting groups
Arm/Group | Total Topiramate Group | Total Placebo Group | Total
Number analyzed (Participants) | 67 | 71 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] — Enrollment was open to participants age 18 to 65 years old
  years | 49.3 (9) | 52.8 (7.4) | 51.07 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 45 | 41 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants] — We collect information about race from participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 4 | 14
    White | 56 | 66 | 122
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Proportion Heavy drinking Days preceding screening visit [Mean (Standard Deviation); unit: Proportion Heavy drinking days] — Proportion of Heavy drinking Days, 90 days preceding the screening visit
  Proportion Heavy drinking days | .67 (.27) | .66 (.27) | .66 (.27)
Location of enrollment [Number; unit: participants] — Connecticut subjects were enrolled at the University of Connecticut and Philadelphia subjects at the University of Pennsylvania.
  participants
    University Of Connecticut | 39 | 37 | 76
    University of Pennsylvania | 28 | 34 | 62
Education [Mean (Standard Deviation); unit: years] — Level of Education measured in years of education.
  years | 15.8 (2.5) | 15.3 (2.5) | 15.5 (2.5)
Marital Status [Number; unit: Number of participants] — Total number married
  Number of participants
    Married | 39 | 45 | 84
    Not married | 28 | 26 | 54
Annual Income [Number; unit: participants] — Annual income measured in categorical amounts
  participants
    Less than $40,000 | 6 | 9 | 15
    $40,000-$79,999 | 14 | 15 | 29
    $80,000 -$119,000 | 18 | 19 | 37
    $120,000 or more | 28 | 28 | 56
    Missing | 1 | 0 | 1
Beck Depression Inventory score [Mean (Standard Deviation); unit: units on a scale] — Total Beck Depression Inventory score The Beck Depression Inventory (BDI), a 21-item self-report measure of depressive symptoms, yields a total score that ranges from 0 to 63, higher scores indicating higher depression (Beck et al. 1961). The BDI is generally regarded as a sensitive self-report measure of depressive symptoms, and will be used to explore the relation between depressive symptoms and response to medication and counseling.
  units on a scale | 6.1 (4.8) | 6.8 (5.3) | 6.48 (5.07)
Proportion of abstinent days [Mean (Standard Deviation); unit: Proportion of abstinent days] — Proportion of abstinent days, 90 days preceding the screening visit.
  Proportion of abstinent days | 0.13 (0.16) | 0.12 (0.15) | 0.12 (0.15)
Short Index of Problems [Mean (Standard Deviation); unit: units on a scale] — The Short Inventory of Problems (SIP). The SIP, a 15-item instrument, yields a total score that ranges from 0 to 45, higher score worse outcomes. The SIP was derived from the Drinker Inventory of Consequences (DrInC), which was developed for use in Project MATCH (Miller and Tonigan 1995). We (Feinn et al. 2003) have found that, like the DrInC, the SIP measures a single factor of alcohol-related problems. Given that it is substantially shorter than the DrInC, we will use the SIP as a measure of alcohol-related consequences.
  units on a scale | 14.9 (8.6) | 15.5 (6.7) | 15.20 (7.6)
Lifetime major depression (M.D.) [Number; unit: # of participants] — Lifetime episode of major depression based on a Structured Clinical Interview for DSM-IV (SCID-I/P) (First et al. 2001). The SCID Module A: Mood Episodes was used to classify patients according to the presence or absence of Lifetime episode of major depression. The SCID-I/P is a procedure designed to determine diagnoses and symptoms according to DSM-IV (American Psychiatric Association 1994).
  # of participants
    Lifetime episode Major Depression | 18 | 22 | 40
    No lifetime Major Depression episode | 49 | 49 | 98
Genotype [Number; unit: Participants]
  CC | 23 | 31 | 54
  AC | 29 | 32 | 61
  AA | 15 | 8 | 23
Mean Daily Alcohol Consumption [Mean (Standard Deviation); unit: Number of SD Drinks per day] | 5.426 (2.019) | 5.207 (1.735) | 5.314 (1.875)

OUTCOME MEASURES:

1. Primary Outcome: Mean Heavy Drinking Days Per Week by Medication Group
Description: Change in the number of heavy drinking days during treatment phase of study. Drinking data were aggregated to the weekly level. The number of days per week of heavy drinking (i.e., four or more drinks in a day for women and five or more drinks in a day for men) and of abstinence were the primary outcomes.
Time Frame: 12 weeks (from initiation to end of treatment)
Population: Intention to treat (ITT)
Measure: Mean (Standard Error); unit: Number of heavy drinking days
Groups:
- Active Med: Topiramate (up to 200 mg orally)
  Medication: Topiramate (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
- Placebo Group: placebo
  placebo: placebo (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
Arm/Group | Active Med | Placebo Group
Number analyzed (Participants) | 67 | 71
Number of heavy drinking days | 1.82 (0.082) | 2.94 (0.091)
Statistical Analysis 1: Comparison: Active Med vs Placebo Group; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Mean Abstinent Days Per Week by Medication Group
Time Frame: 12 weeks
Population: Intention to treat (ITT).
Measure: Mean (Standard Error); unit: Mean abstinent days per week
Arm/Group | Active Med | Placebo Group
Number analyzed (Participants) | 67 | 71
Mean abstinent days per week | 2.00 (0.085) | 1.36 (0.065)
Statistical Analysis 1: Comparison: Active Med vs Placebo Group; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

3. Secondary Outcome: Mean Daily Alcohol Consumption
Time Frame: 12 weeks (from initiation to end of treatment); 3- and 6-months post-treatment
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: Standard Drinks per day
Groups:
- 3 Month Post Treatment Topiramate Group; 3 Month Post Treatment Placebo Group: Mean Standard Drinks Per Day, 3 months post treatment
- 6 Month Post Treatment Topiramate Group; 6 Month Post Treatment Placebo Group: Mean Standard Drinks Per Day, 6 months post treatment
Arm/Group | Total Topiramate Group | Total Placebo Group | 3 Month Post Treatment Topiramate Group | 3 Month Post Treatment Placebo Group | 6 Month Post Treatment Topiramate Group | 6 Month Post Treatment Placebo Group
Number analyzed (Participants) | 67 | 71 | 60 | 63 | 59 | 59
Standard Drinks per day | 2.9859 (2.01983) | 3.5523 (1.59254) | 2.6129 (1.84037) | 2.7560 (1.92299) | 2.6448 (2.00703) | 2.8377 (1.96230)

4. Secondary Outcome: Mean Heavy Drinking Days Per Week by Medication Group and rs2832407 Genotype
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Error); unit: Mean Heavy Drinking Days Per Week
Groups:
- Topiramate CC Genotype; Topiramate AC Genotype; Topiramate AA Genotype: topiramate (up to 200 mg orally)
  topiramate: up to 200mg/day orally (over 12 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
- Placebo CC Genotype; Placebo AC Genotype; Placebo AA Genotype: placebo
  placebo: placebo (12 weeks during which the dosage of study medication is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
Arm/Group | Topiramate CC Genotype | Placebo CC Genotype | Topiramate AC Genotype | Placebo AC Genotype | Topiramate AA Genotype | Placebo AA Genotype
Number analyzed (Participants) | 21 | 30 | 24 | 29 | 11 | 7
Mean Heavy Drinking Days Per Week | 1.28 (0.131) | 3.49 (0.141) | 2.30 (0.130) | 2.72 (0.129) | 1.8 (0.163) | 1.54 (0.211)
Statistical Analysis 1: Comparison: Topiramate CC Genotype vs Placebo CC Genotype vs Topiramate AC Genotype vs Placebo AC Genotype vs Topiramate AA Genotype vs Placebo AA Genotype; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis

5. Secondary Outcome: Mean Abstinent Days Per Week by Medication Group and rs2832407 Genotype
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Error); unit: Mean Abstinent Days Per Week
Arm/Group | Topiramate CC Genotype | Placebo CC Genotype | Topiramate AC Genotype | Placebo AC Genotype | Topiramate AA Genotype | Placebo AA Genotype
Number analyzed (Participants) | 21 | 30 | 24 | 29 | 11 | 7
Mean Abstinent Days Per Week | 2.41 (0.148) | 1.02 (0.090) | 1.51 (0.119) | 1.44 (0.095) | 2.26 (0.186) | 2.49 (0.227)
Statistical Analysis 1: Comparison: Topiramate CC Genotype vs Placebo CC Genotype vs Topiramate AC Genotype vs Placebo AC Genotype vs Topiramate AA Genotype vs Placebo AA Genotype; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis

6. Secondary Outcome: Severity of Alcohol-related Problems at End of Treatment
Description: The Short Inventory of Problems (SIP). The SIP, a 15-item instrument, yields a total score that ranges from 0 to 45, higher score indicating higher levels of drinking problems. The SIP was derived from the Drinker Inventory of Consequences (DrInC), which was developed for use in Project MATCH (Miller and Tonigan 1995). We (Feinn et al. 2003) have found that, like the DrInC, the SIP measures a single factor of alcohol-related problems. Given that it is substantially shorter than the DrInC, we will use the SIP as a measure of alcohol-related consequences.
Time Frame: 12 weeks (from intiation to end of treatment)
Population: Subject were measured at Baseline and Endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Med | Placebo
Number analyzed (Participants) | 67 | 71
units on a scale | 7.0 (7.2) | 11.1 (7.5)
Statistical Analysis 1: Comparison: Active Med vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

7. Secondary Outcome: Gamma-glutamyl Transferase (GGT) at Midpoint
Description: Gamma-glutamyl transferase (GGT) is a liver enzyme biochemical measure used to detect liver health and function and alcohol consumption. GGT is a very sensitive measure than can change very quickly compared to other biochemical markers.
Time Frame: 6 weeks (from initiation to midpoint)
Population: Subjects were measured at midpoint.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Active Med | Placebo
Number analyzed (Participants) | 59 | 64
IU/L | 37.6 (36.7) | 50.1 (64.8)
Statistical Analysis 1: Comparison: Active Med vs Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis

8. Secondary Outcome: Gamma-glutamyl Transferase (GGT) at End of Treatment
Description: as for outcome 7
Time Frame: 12 weeks (from initiation to end of treatment)
Population: ITT
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Active Med | Placebo Group
Number analyzed (Participants) | 58 | 63
IU/L | 36.3 (40.2) | 47.9 (52.1)
Statistical Analysis 1: Comparison: Active Med vs Placebo Group; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of enrollment, throughout the 12 week treatment phase and 6 month followup phase of the study.
Groups:
- Topiramate Group: topiramate (up to 200 mg orally)
  topiramate: up to 200mg/day orally (over 12 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
Arm/Group | Topiramate Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/71
Other Adverse Events (participants affected / at risk) | 36/67 | 16/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate Group (N=67) | Placebo Group (N=71)
Numbness/Tingling (General disorders) | 36 | 10
Change in taste (General disorders) | 25 | 6
Tireness/Sleepiness (General disorders) | 18 | 16
Difficulty with memory (General disorders) | 16 | 16
Loss of appetite (General disorders) | 16 | 2
Headache (General disorders) | 15 | 14
Diarrehea (General disorders) | 14 | 10
Weight loss (General disorders) | 13 | 2
Difficulty Concentrating (General disorders) | 12 | 4
Dry Mouth (General disorders) | 11 | 4
Nausea (General disorders) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes